CLINICAL TRIAL: NCT04378465
Title: Enhanced Recovery Program in Laparoscopic Colorectal Surgery: an Observational Controlled Trial
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Other Study IDs: 52-2011
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Surgery; Recovery of Function
Keywords: Laparoscopy; Enhanced Recovery After Surgery; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERP group: A prospective series of consecutive patients undergoing elective colorectal surgery completing a standardized Enhanced Recovery Program (ERP) protocol at the S. Anna University Hospital in Ferrara (Italy) in 2013-2015
  Interventions: Other: Enhanced Recovery Program (ERP)
- Non-ERP group: A retrospective series of consecutive patients operated at the same hospital (S. Anna University Hospital in Ferrara), in the same period of time (2013-2015), but with a traditional perioperative care protocol.

INTERVENTIONS:
Other: Enhanced Recovery Program (ERP) — An evidence-based perioperative care approach, involving a multidisciplinary team work including surgeons, anaesthesiologists, dieticians, and nurses, which aim to reduce the surgical stress and metabolic responses as well as organ dysfunction, thus leading to a faster recovery after surgery
  Groups: ERP group

SUMMARY:
Background: A few randomized clinical trials and meta-analysis provide evidence for enhanced recovery programs (ERPs) in colorectal surgery. Most of the evidence, however, relies on non-randomized controlled studies that have control groups being either historical or operated on at different facilities. The aim of this study was to compare a prospective series of patients undergoing elective colorectal surgery according to ERPs, with a coeval retrospective series of patients undergoing elective colorectal surgery in a different ward at the same hospital.

The primary outcome was hospital length of stay, which was used as a proxy of functional recovery. Secondary outcomes included: postoperative complications, readmission rate, mortality, and adherence to the protocol.

Materials and Methods: A prospective series of consecutive patients (N = 100) undergoing elective colorectal resection completing a standardized ERP in 2013-2015 (ERP Group) will be compared to patients (N = 100) operated at the same institution in the same period with a traditional perioperative care protocol (Non-ERP group). Despite different surgeons and ward nurses, the two groups shared the same anaesthesiologists and were located in separate wards. The exclusion criteria were: >80 years old, ASA score of IV, a stage IV TNM, and diagnosis of inflammatory bowel disease.

DETAILED DESCRIPTION:
1. Introduction

   One of the most important achievements in modern surgery is the implementation in perioperative care of Enhanced Recovery Programs (ERPs), pioneered by Henrik Kehlet in the mid-1990s [1]. ERP is an evidence-based perioperative care approach, involving a multidisciplinary team work including surgeons, anaesthesiologists, dieticians, and nurses, which aim to reduce the surgical stress and metabolic responses as well as organ dysfunction, thus leading to a faster recovery after surgery [2].

   Such a team works with a multimodal approach to perioperative care, sharing all the endpoints of management throughout the perioperative phases, and acting in close relationship with the patient along his/her "journey in hospital". In other words, each perioperative phase comprises several core items based on solid scientific evidence that are delivered by different professionals in different parts of the hospital [2].

   A few randomized clinical trials and meta-analysis provide evidence in the literature for the benefits of ERPs in colorectal surgery [3-6]. Most non-randomized controlled studies have compared patients undergoing colorectal enhanced recovery surgery with controls being either historical groups or patients operated on at different hospitals [7-9].

   In a previous investigation, the investigators showed the benefits of implementing an ERP in elective colorectal surgery by comparing a prospective series of 100 patients operated on receiving enhanced recovery care (ERP group), with a retrospective cohort of 100 patients operated on by the same professionals at the same institution before the introduction of the ERP (Pre-ERP group) [10].

   The present study aims to investigate the differences between a prospective series of patients undergoing elective colorectal surgery following an ERP and a retrospective cohort of patients operated on with traditional perioperative care in the same period by a different team of surgeons and hospitalized in a different ward of the same hospital.
2. Materials and Methods

The study was designed as a prospective cohort with retrospective coeval control. A prospective series of 100 consecutive patients undergoing elective colorectal surgery completing a standardized ERP protocol at the S. Anna University Hospital in Ferrara (Italy) in 2013-2015 (ERP group), was compared to a retrospective series of 100 consecutive patients operated at the same hospital, in the same period of time, but with a traditional perioperative care protocol (Non-ERP group). Despite different surgeons and ward nurses, the two groups of patients shared the same anaesthesiologists and were located in two separate wards.

In 2012 the enhanced recovery team was assembled, the ERP protocol was built up, according to the fast-track protocol proposed by Kehlet and Wilmore [11], and periodical audits were then performed. Eligible for this study were all patients between 18 and 80 years old scheduled for elective colorectal resection. Exclusion criteria in both study groups were: age > 80 years old, American Society of Anaesthesia (ASA) score IV, TNM stage IV, and diagnosis of inflammatory bowel disease. Discharging criteria were also the same for both groups: 1) free oral diet, 2) complete intestinal function recovery (passage of flatus and stool), 3) dynamic pain control (Numerical Rate Scale - NRS ≤ 3) by oral analgesia, 4) independent walking, 5) no signs of infection [10].

The study protocol was approved by the local Ethics Committee (Ethical Committee for Human Subject Research study number 52-2011), it complies with the Declaration of Helsinki, and all patients provided written informed consent The primary outcome of this study was the length of stay (LoS) in the hospital, adopted as a proxy of functional recovery. Secondary outcomes were: postoperative complications, readmission rate, mortality, and adherence to the protocol.

All complications were recorded until 30 days after surgery, as well as mortality and hospital readmission. To evaluate adherence to the protocol, all ERP items were prospectively collected, recorded and checked by an independent observer using a detailed care program for each postoperative day. The grading of complications was defined according to a validated classification [12].

Data were collected prospectively for patients in the ERP group and retrieved from a prospectively maintained database for those in the Non-ERP group.

Surgery was preferably performed by laparoscopy, but alternative approaches were allowed and discussed with patients. A converted laparoscopy was defined as an unplanned extension of the surgical incision (either a median or a transverse suprapubic incision). All operations were performed by surgeons experienced in colorectal surgery and advanced laparoscopy (CVF, GA).

2.1 ERP Group Patients received extensive preoperative counselling about protocol items, all phases of perioperative care, and discharge criteria, along with an illustrated booklet conceived by the multidisciplinary team. The patients were motivated to adhere to protocol items by members of the team throughout the preoperative and postoperative phases and were informed about the daily objectives to be achieved. Incentive spirometers were provided preoperatively and patients were instructed for perioperative breathing exercises.

A normal meal was allowed on the day before surgery; a carbohydrate loaded drink was prescribed in the evening (100 grams of maltodextrin in 800 ml liquid drink) and at least two hours (50 grams of maltodextrin in 400 ml liquid drink) before surgery. No patient was prescribed mechanical bowel preparation.

The nasogastric tube (NGT) and bladder catheter were removed at the end of the procedure and within the second postoperative day [13], respectively, whereas abdominal drains were selectively used.

Postoperative pain control was achieved with thoracic epidural analgesia within the first three postoperative days and with Nonsteroidal Anti-Inflammatory Drugs (NSAIDs) or paracetamol thereafter. Resumption of liquid and solid diets and discontinuation of intravenous fluids were all achieved within the first and the second postoperative day. Patients were out of bed on postoperative day one and encouraged by nurses to deambulate according to a predefined schedule.

The anaesthetic protocol was standardized as previously described elsewhere [10]. In brief, a blended anaesthesia was performed with short-acting anaesthetic agents and mid-thoracic epidural intraoperative analgesia. Attention was put on maintaining normothermia with forced air warming devices during surgical procedures and a multimodal approach to prevent PostOperative Nausea and Vomiting (PONV) was pursued. Intravenous fluid overload was avoided.

2.2 Non-ERP Group Patients were treated according to traditional perioperative care principles in use at the institution. Specifically, on the day before surgery patients fasted from midnight, received no carbohydrate loaded drink, and performed a mechanical bowel preparation.

An opioid-based anaesthesia with or without thoracic epidural was used, while postoperative pain control was achieved by intravenous opioids, thoracic epidural or NSAIDs.

The NGT was removed at the restoration of intestinal activity when oral feeding was resumed, while the abdominal drain was removed at bowel movements.

No predefined schedule was followed for patients' mobilization and the bladder catheter was removed at full mobilization and after discontinuation of intravenous fluids.

Patients received no daily goal assignments or specific preoperative counselling.

In order to determine in between groups perioperative care differences, an independent observer reviewed the medical charts of all patients to evaluate the adherence to the 21 protocol items.

2.3 Statistical Analysis Clinical parameters were expressed as median (interquartile range - IQR 25-75) and mean ± standard deviation according to distribution assessed by Shapiro-Wilk test. Categorical data were presented as numbers. Clinical and pathological variables were analysed with Chi-square, t-student, and Mann-Whitney tests as appropriate. The Kaplan-Meier test method and Log-Rank test were used to compare duration of surgical operation, time to functional recovery and hospital LoS between groups. A P value of less than 0.05 was considered statistically significant. Statistical analysis was performed with IBM SPSS Statistics for Windows, Version 24.0 (IBM Corp. Armonk, NY: IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing elective colorectal resection at the S. Anna University Hospital in Ferrara (Italy)

Exclusion Criteria:

* age >80 years old,
* American Society of Anesthesia (ASA) score IV,
* TNM stage IV,
* inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective colorectal resection at the S. Anna University Hospital in Ferrara (Italy) between 2013-2015 (ERP group vs Non-ERP group)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Postoperative Hospital Length Of Stay (LOS) | Within 10 days from date of surgical operation
  The postoperative hospital LOS, proxy of functional recovery, is defined as the number of days from the date of surgical operation to the date of hospital. Patients in both study groups wil be discharged from the hospital upon reaching all predefined discharged criteria. For the ERP group it is estimated a 4 to 5-day hospital LOS according to the protocol, while in the traditional group an 8 to 10-day hospital stay is expected.

SECONDARY OUTCOMES:
Morbidity | Within 30 days from date of surgical operation
  Postoperative complications
Mortality | Within 30 days from date of surgical operation
  Postoperative mortality rate
30-day readmission | Within 30 days from date of surgical operation
  30-day readmission rate to the hospital
Adherence to the ERP protocol | Within 10 days from date of surgical operation
  The ERP protocol includes 21 items; the adherence to the items will be evaluated for each patient in the postoperative period. Then, the adherence rate will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo V Feo, MD, Principal Investigator — University Hospital of Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Wang Q, Suo J, Jiang J, Wang C, Zhao YQ, Cao X. Effectiveness of fast-track rehabilitation vs conventional care in laparoscopic colorectal resection for elderly patients: a randomized trial. Colorectal Dis. 2012 Aug;14(8):1009-13. doi: 10.1111/j.1463-1318.2011.02855.x. PMID 21985126
- [Background] Lee TG, Kang SB, Kim DW, Hong S, Heo SC, Park KJ. Comparison of early mobilization and diet rehabilitation program with conventional care after laparoscopic colon surgery: a prospective randomized controlled trial. Dis Colon Rectum. 2011 Jan;54(1):21-8. doi: 10.1007/DCR.0b013e3181fcdb3e. PMID 21160309
- [Background] Serclova Z, Dytrych P, Marvan J, Nova K, Hankeova Z, Ryska O, Slegrova Z, Buresova L, Travnikova L, Antos F. Fast-track in open intestinal surgery: prospective randomized study (Clinical Trials Gov Identifier no. NCT00123456). Clin Nutr. 2009 Dec;28(6):618-24. doi: 10.1016/j.clnu.2009.05.009. Epub 2009 Jun 17. PMID 19535182
- [Background] Zhao JH, Sun JX, Gao P, Chen XW, Song YX, Huang XZ, Xu HM, Wang ZN. Fast-track surgery versus traditional perioperative care in laparoscopic colorectal cancer surgery: a meta-analysis. BMC Cancer. 2014 Aug 23;14:607. doi: 10.1186/1471-2407-14-607. PMID 25148902
- [Background] Pedziwiatr M, Kisialeuski M, Wierdak M, Stanek M, Natkaniec M, Matlok M, Major P, Malczak P, Budzynski A. Early implementation of Enhanced Recovery After Surgery (ERAS(R)) protocol - Compliance improves outcomes: A prospective cohort study. Int J Surg. 2015 Sep;21:75-81. doi: 10.1016/j.ijsu.2015.06.087. Epub 2015 Jul 29. PMID 26231994
- [Background] Depalma N, Cassini D, Grieco M, Barbieri V, Altamura A, Manoochehri F, Viola M, Baldazzi G. Feasibility of a tailored ERAS programme in octogenarian patients undergoing minimally invasive surgery for colorectal cancer. Aging Clin Exp Res. 2020 Feb;32(2):265-273. doi: 10.1007/s40520-019-01195-6. Epub 2019 Apr 13. PMID 30982218
- [Background] Aarts MA, Rotstein OD, Pearsall EA, Victor JC, Okrainec A, McKenzie M, McCluskey SA, Conn LG, McLeod RS; iERAS group. Postoperative ERAS Interventions Have the Greatest Impact on Optimal Recovery: Experience With Implementation of ERAS Across Multiple Hospitals. Ann Surg. 2018 Jun;267(6):992-997. doi: 10.1097/SLA.0000000000002632. PMID 29303803
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Zaouter C, Kaneva P, Carli F. Less urinary tract infection by earlier removal of bladder catheter in surgical patients receiving thoracic epidural analgesia. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):542-8. doi: 10.1097/aap.0b013e3181ae9fac. PMID 19916208
- [Result] Portinari M, Ascanelli S, Targa S, Dos Santos Valgode EM, Bonvento B, Vagnoni E, Camerani S, Verri M, Volta CA, Feo CV. Impact of a colorectal enhanced recovery program implementation on clinical outcomes and institutional costs: A prospective cohort study with retrospective control. Int J Surg. 2018 May;53:206-213. doi: 10.1016/j.ijsu.2018.03.005. Epub 2018 Mar 13. PMID 29548700